CLINICAL TRIAL: NCT03050788
Title: Smartphone Confocal Microscopy for Diagnosing Kaposi's Sarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Infectious Diseases Institute, Uganda (Other)
Responsible Party: Principal Investigator, Dongkyun Kang, Assistant Professor of Dermatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016P002672
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Kaposi Sarcoma
Keywords: Smartphone confocal microscopy; Kaposi Sarcoma; Point of care diagnosis
MeSH Terms: conditions — Sarcoma, Kaposi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smartphone confocal microscopy imaging (Experimental): Subject's skin lesion will be imaged with the smartphone confocal microscopy.
  Interventions: Device: Smartphone confocal microscopy

INTERVENTIONS:
Device: Smartphone confocal microscopy — Imaging of skin lesion using the smartphone confocal microscopy

SUMMARY:
The investigators propose to evaluate a novel diagnostic approach for Kaposi's sarcoma (KS) that may be eventually deployed with portable, point-of-care techniques. This approach features confocal microscopy. The investigators will compare this new approach with the gold standard of histology from a traditional skin punch biopsy (which is standard of care) to determine the sensitivity and specificity of portable confocal microscopy in diagnosing KS.

DETAILED DESCRIPTION:
The investigators will perform a cross-sectional study of 500 patients in routine clinical care settings who are suspected to have KS on clinical grounds and for whom skin punch biopsy and histopathological examination is indicated as part of standard of care. Patients will be evaluated with both the gold standard for diagnosis of KS (skin punch biopsy followed by histopathology) and portable confocal microscopy.

ELIGIBILITY:
Inclusion Criteria:

i. ≥ 18 years old ii. Clinically suspected KS iii. Presence of suspected KS lesions in areas which are considered safe to biopsy by the Ugandan providers, which means all areas of the skin except for the mouth and eye.

Exclusion Criteria:

i. Presence of suspected KS lesions exclusively on the mouth or eye unless clinical specialists trained in biopsy of the mouth or eye are available locally to biopsy the mouth or eye. Oral and eye sites would typically only be biopsied when clinical diagnosis has proved to be problematic and definitive diagnosis is needed to inform a treatment plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of diagnosing Kaposi sarcoma using the smartphone confocal microscopy | Approximately 20 minutes (10 minutes for in vivo imaging)
  Confocal microscopy images obtained from the skin lesion will be compared with the corresponding histologic images. Diagnostic accuracy will be tested. No clinical decisions will be made based on confocal microscopy images.

CONTACTS AND LOCATIONS:
Overall Officials: Dongkyun Kang, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No